CLINICAL TRIAL: NCT01832766
Title: The Effects of Cannabis Use in People With Schizophrenia on Clinical, Neuropsychological and Physiological Phenotypes
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Unable to find subjects with schizophrenia that were using only cannabis
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Alliance for Research on Schizophrenia and Depression (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple
Other Study IDs: 05-0359
Record Dates: First submitted 2013-03-25; First posted 2013-04-16 (Estimated); Results first posted 2015-09-21 (Estimated); Last update posted 2015-09-21 (Estimated); Status verified 2015-08

CONDITIONS: Schizophrenia
Keywords: schizophrenia; dronabinol; P50; cannabis; memory; symptoms
MeSH Terms: conditions — Schizophrenia; Marijuana Abuse | interventions — Dronabinol; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- dronabinol (Active Comparator): dronabinol 10 mg one capsule by mouth at 8:00 a.m.
  Interventions: Drug: Dronabinol
- sugar pill (Placebo Comparator): one capsule given by mouth at 8:00 a.m.
  Interventions: Other: Placebo Comparator

INTERVENTIONS:
Drug: Dronabinol — dronabinol 10 mg one capsule by mouth at 8:00 a.m.
  Other Names: Marinol
  Arms: dronabinol
Other: Placebo Comparator — one capsule given by mouth at 8:00 a.m.
  Other Names: Sugar Pill
  Arms: sugar pill

SUMMARY:
Approximately 25% of people with schizophrenia abuse marijuana. These people may be using marijuana to self-medicate symptoms such as hallucinations (hearing or seeing things that are not heard or seen by others) or delusions (false beliefs i.e. people are harassing or persecuting them) or the depressed and anxious feelings brought on by these symptoms. Currently, it is unknown whether marijuana makes schizophrenia better or worse. Marijuana intoxication in people without schizophrenia generally causes decreased recall of words, may decrease reaction time and decrease inhibition. Additionally, marijuana may cause distractibility as demonstrated by difficulty keeping their eyes on a moving target and difficulty inhibiting their response to repetitive tones. However, marijuana may have different effects in schizophrenia. Receptors for cannabis (marijuana) are concentrated in the brain and maladjustment of the cannabinoid system may be associated with the difficulty in thinking found in schizophrenia. The proposed research project examines if clinical symptoms, learning, memory, inhibition and distractibility are improved or made worse by the acute ingestion of tetrahydrocannabinol (THC).

DETAILED DESCRIPTION:
The trial will be a double two period (visit) blind cross-over trial with one arm dronabinol 10 mg one arm a placebo control. The order of doses and placebo will be randomized with the restriction that half of the subjects will receive each order. This counterbalances possible visit effects or learning effects associated with the visits. The use of an oral cannabis analog is not equivalent to smoking as the onset of action is slower. This is why people who use dronabinol for chronic pain prefer to smoke cannabis. There is no "high" associated with dronabinol. However, the active ingredients are the same, THC, which will have similar effects on the cannabinoid 1 receptor. Ethically, we did not feel we could ask people to smoke cannabis on one day of study. Subjects will present to the GCRC at 5:00 p.m. They will abstain from use of cannabis overnight. The following morning, at 8:00 a.m., the subject will provide a urine sample for a toxicology screen and a blood sample for quantitative THC levels. They will then be administered either 10 mg of dronabinol or an identical placebo on an alternate day. The subject will then have a baseline assessment of clinical positive and negative symptoms measured by the Brief Psychiatric Rating Scale (BPRS). The majority (70-90%) of people with schizophrenia smoke cigarettes. Thus, it is likely that in this population that smokes cannabis, 100% will also be cigarette smokers. The effects of nicotine via cigarette smoking on the endophenotypes studied is an acute effect, with a peak at about 5 minutes. To preclude nicotine effects on endophenotypes, we have the patient not smoke for 20 minutes prior to and during testing. Nicotine is quickly removed from the body when inhaled and its effects wear off within 20 minutes. Two hours after administration, the subject will perform the following tests: P50 auditory evoked potential- the recording will consist of the presentation of 5 sets of 16 click pairs with an intrapair interval of 500 ms heard through headphones with a 3-minute rest between sets. Brain wave responses will be recorded; neurocognitive assessment-the California Verbal Learning Test will measure verbal memory and the Stroop will measure inhibition; clinical symptom assessment- The BPRS will again be administered measure positive and negative symptoms; and a blood sample will be collected for quantitative THC levels. They will then be escorted by a Clinical Research Center nurse over to a laboratory at Colorado Psychiatric Hospital to perform smooth pursuit eye movements In performing smooth pursuit eye movements, they will watch a dot moving across a computer screen while infrared sensors that are placed just in front of their eyes record their eye movements. Each subject performs 3 trials of one minute each, with 2 minutes rest between each recording. Subjects will be reassessed by the BPRS for drug exacerbation of symptoms, will have vitals, will be checked for adverse effects, will perform a sobriety test (the standard test used in roadside testing i.e. walking a straight line and finger to nose testing) which will be assessed by Dr. Olincy, who is experienced in assessing sobriety, to assure that the patient is not acutely intoxicated and able to perform normal functions that require coordination. If they fail the sobriety test, they will be asked to remain in the (General Clinical Research Center (GCRC) until they can pass the sobriety test. Otherwise, they will then will be discharged at 5:00 p.m. Transportation to and from the GCRC will be by a provided cab service. Subjects will be randomized in blocks of 4 or 6 to the order in which they receive placebo or dronabinol. The interval between the two days of testing will be 1 week.

ELIGIBILITY:
Inclusion Criteria:

* Male and females
* 18 and 50 years of age
* Diagnosis of schizophrenia
* Chronic cannabis users who have used for at least 1 year
* Using cannabis at least once weekly
* Currently being treated with antipsychotic medication
* Must be on a the same dose of antipsychotic medication for at least 3 months.
* Females of childbearing potential must use an adequate form of birth control while participating.
* Participants will be required to have blood pressures greater than 90/60 and less than 140/90.

Exclusion Criteria:

* Use of illicit drugs other than cannabis
* Any psychiatric hospitalizations within 3 months
* pregnancy in females
* taking clozapine

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2005-06; Primary Completion 2010-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lynn Johnson, Pharm D, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Denver, Aurora, Colorado, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Age-eligible participants were recruited from May 2005 to May 2010 and were recruited from local mental health centers.
Pre-assignment Details: 14 recruited; 14 screened: 1 excluded (did not meet inclusion criteria)
Groups:
- Dronabinol 10 mg First Then Placebo: dronabinol 10 mg given oral one dose in first intervention period then 1 week washout period and then placebo given oral in one dose in second intervention period
- Placebo First Then 10 mg Dronabinol: identical capsule given orally once in first intervention period then 1 week washout period then dronabinol 10 mg given orally once in second intervention period
Period: First Intervention
Arm/Group | Dronabinol 10 mg First Then Placebo | Placebo First Then 10 mg Dronabinol
Started | 7 | 6
Completed | 7 | 6 (one participant did not return for cross over visit)
Not Completed | 0 | 0
Period: Washout
Arm/Group | Dronabinol 10 mg First Then Placebo | Placebo First Then 10 mg Dronabinol
Started | 7 | 6
Completed | 7 | 5
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1
Period: Second Intervention
Arm/Group | Dronabinol 10 mg First Then Placebo | Placebo First Then 10 mg Dronabinol
Started | 7 | 5
Completed | 7 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Entire Study Population: includes groups randomized to receive placebo first or dronabinol 10 mg first
Arm/Group | Entire Study Population
Number analyzed (Participants) | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 32 (11.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 10
Region of Enrollment [Number; unit: participants]
  United States | 13

OUTCOME MEASURES:

1. Primary Outcome: P50 Auditory Evoked Potential
Description: electrophysiological measure of ability to filter extraneous stimuli measured as the amplitude of the evoked response to the second auditory stimulus divided by the amplitude of the evoked response to the first auditory stimulus in mV.
Time Frame: 2 hours after drug administration
Population: One participant did not complete the treatment or the placebo arm (crossover study design).
Measure: Mean (Standard Deviation); unit: test to conditioning ratio
Groups:
- Dronabinol: dronabinol 10 mg given oral one dose
- Placebo: identical capsule given once
Arm/Group | Dronabinol | Placebo
Number analyzed (Participants) | 12 | 12
test to conditioning ratio | .62 (.69) | .52 (.43)

2. Secondary Outcome: California Verbal Learning Test Change at 2 Hours From Baseline
Description: ability to remember a list of words given 5 trials. Number of words remembered is normalized to a schizophrenia population and average scores are calculated with age correction. The normal T-score is 50 and scores greater than 50 correspond with greater ability to remember words as compared to a schizophrenia population norm.
Time Frame: 2 hours after drug administration
Population: One participant did not complete the treatment or the placebo arm (crossover study design).
Measure: Mean (Standard Deviation); unit: T scores
Arm/Group | Dronabinol | Placebo
Number analyzed (Participants) | 12 | 12
T scores | -.5 (1.92) | -.77 (1.19)

3. Other Pre Specified Outcome: Brief Psychiatric Rating Scale Change From Baseline at 1 Hour
Description: Measures psychiatric symptoms. Each item is scored from 1-7. Positive symptoms are calculated from sum of scores on hallucinatory behavior, unusual thought content and conceptual disorganization. Thus, the range of Total Positive Symptoms can be from a score of 3-21 .The higher the score, the more severe the symptom. Negative symptoms have been calculated from sum of blunted affect, emotional withdrawal and motor retardation. The range of Total Negative Symptoms can be from a score of 3-21. The higher the score, the more severe the symptoms. As this is a difference from baseline, there can be either negative or positive results as the subjects can either be better than baseline (positive score) or worse than baseline (negative score).
Time Frame: at 1 hour after drug administration
Population: One participant did not complete the treatment or the placebo arm (crossover study design).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Dronabinol | Placebo
Number analyzed (Participants) | 12 | 12
units on a scale | 3.73 (1.1) | 3.18 (.6)

ADVERSE EVENTS:
Arm/Group | Dronabinol | Placebo
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 0/13 | 0/13

LIMITATIONS AND CAVEATS:
early termination as recruitment of subjects with only cannabis use was difficult leading to small number of subjects analyzed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No